CLINICAL TRIAL: NCT03211520
Title: Magnetic Resonance Imaging:A Window to Anthracycline Toxicity
Status: Completed | Type: Observational
Sponsor: Connecticut Children's Medical Center (Other)
Responsible Party: Principal Investigator, Tiffany Ruiz, Cardio-oncology nurse program manager, Connecticut Children's Medical Center
Other Study IDs: 10-066
Record Dates: First submitted 2017-02-13; First posted 2017-07-07 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Cardiac Complications
Keywords: Cancer treatment; Anthracyclines; Cardiac MRI

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Pending
Oversight: Data Monitoring Committee: No

SUMMARY:
The study is being conducted to see which cardiac tests that monitor how the heart functions during and after treatment with anthracyclines are most effective. This study will assess a new way to check the heart function of children during and after cancer treatment. Currently, doctors use echocardiograms (heart ultrasound) to see how the heart is working. Echocardiograms are currently being done as part of standard of care prior to giving anthracycline chemotherapy doses and if any cardiac problems are suspected. The new method involves Cardiac Magnetic Resonance Imagining (CMRI) and a blood tests for certain biomarkers for heart health: High sensitivity troponin, Caspase, C-reactive Protein (CRP), ventricular derived B-type natriuretic peptide (BNP), Matrix Metalloproteinases (MMPs), Tissue inhibitors of metalloproteinases (TIMPs), C terminal propeptide of type I procollagen (PICP), C terminal telopeptide of collagen type I (CITP), Troponin I, and Bone Alkaline Phosphatase. The purpose of this study is to find out if CMRI and blood tests help us to find heart problems earlier, before they are detected by echocardiograms.

DETAILED DESCRIPTION:
This is a pilot study with a descriptive study design.

Anthracycline induced late onset cardiotoxicity, defined in terms of abnormal findings on echocardiography, has been reported to occur in 57% of childhood cancer survivors. Serial monitoring of cardiac function by means of echocardiography detects cardiac toxicity only when many of the cardiomyocytes have already been damaged. Given the lack of evidence to support the reliability of serum markers of cardiotoxicity, many recommend modifying the dose of anthracyclines only when there is objective evidence of myocardial dysfunction by echocardiograph. This approach could be responsible for the increasing frequency of dilated cardiomyopathy occurring 10-15 years after treatment. Non invasive imaging methods are thus critically needed to more precisely detect cardiotoxic changes in children receiving anthracyclines. CMRI has become the gold standard for the assessment and quantification of ventricular volumes, myocardial mass and global and regional wall function. CMRI also allows morphologic analysis of the myocardium as well as detection and characterization of pathological myocardium. In this study, the investigator therefore proposes to use serial MRI parameters in conjunction with a battery of serologic markers, obtained at intervals determined by cumulative anthracycline dose, to monitor changes in systolic function during chemotherapy and one year after the end of chemotherapy. The investigator will use a combination of a serum cardiac biomarker of inflammation (CRP), myocyte injury (Troponin, Caspases), heart failure (BNP), and extracellular matrix remodeling (PICP, CITP, Bone Alkaline Phosphatase, MMPs, TIMPs). The investigator will then correlate these findings with CMRI parameters of myocyte dysfunction. Results will be compared with standard echocardiography. The investigator predict that CMRI is a better indicator of early anthracycline cardiotoxicity in children with solid tumors and hematologic malignancies.

Patients who are of age 9 years of age or older, newly diagnosed with a malignancy that is anticipated to receive high dose anthracyclines as part of their chemotherapy (such as but not limited to solid tumors, high risk Acute Lymphocytic Leukemia, Acute Myelogenous Leukemia, and lymphomas) will be invited to participate in the study.

Specific Aim 1: To use CMRI to detect occult asymptomatic cardiotoxicity over time and in relation to cumulative dose among pediatric cancer patients treated with anthracyclines.

Specific Aim 2: To quantitate serologic biomarker profile for several functional pathways including the inflammatory cascade, MMP/TIMP remodeling pathways, signaling, cell viability and growth domains over time and in relation to cumulative dose among pediatric cancer patients treated with anthracyclines.

Specific Aim 3: To compare changes over time detected by CMRI and serologic markers of cardiac toxicity to echocardiographic indices of systolic and diastolic function and determine their ability alone or in combination to predict freedom from left ventricular dysfunction defined as change in ejection fraction at one year post chemotherapy.

These aims will test the hypothesis that CMR imaging and serologic biomarkers of inflammation, apoptosis and progressive extracellular matrix remodeling will precede echocardiographic indices of systolic and diastolic function among children receiving high dose anthracyclines as part of their chemotherapy protocol.

Study Outcome Measures

Myocardial edema in the acute phase measured by the following parameters:

* Increased myocardial mass.
* Focal areas of high signal intensity T2 weighted spin echo imaging and myocardial delayed enhancement. Significant enhancement will be defined as signal intensity increases of greater than two standard deviations above the mean value of remote normal myocardium.
* Increased myocardial T2 relaxation time in the myocardium compared to baseline as measured by T2 mapping technique
* Changes in myocardial T1 relaxation time in the myocardium pre and post-contrast compared to baseline as measured by T1 mapping technique (Modified Look-Locker inversion recovery (MOLLI). Myocardial T1 (msc).
* Decrease in myocardial strain and strain rate compared to baseline calculations: Mid wall left ventricular circumferential strain (ECC), Maximum longitudinal left ventricular strain (ELL).
* Decrease in myocardial T2* indicative of presence of Iron in the myocardium (reflecting anthracycline-Fe complexes)(ms).
* The following markers were measured: Matrix/Fibrosis pathway:

Plasma levels of MMPs (all soluble MMP types) and TIMPs (all 4 TIMPs); Inflammatory domain: cytokines (TNFα, interleukins, interferon gamma (IFNG), TGF β2, TGF βII)),cytokine receptors (sTNF RI, sTNF RII, sSt2, sgp130, siL1-RII/sCD121b, siL-2Rα/CD25, siL-4R, siL-6R, Endoglin); Signaling pathway: growth factors (GDP-15, GCSF, VEGF, sVEGFR2 TGFβ1, IGF-1;). Changes in regional myocardial function and elevation of serologic markers may predict freedom from left ventricular dysfunction defined as ejection fraction ≥55% at 1 year.

The following tests and procedures will be done for this study:

1. CMRI tests
2. Blood tests
3. Echocardiograms

These tests noted above will be done:

1. Prior to or at before the cum dose of anthracyclines = 60 mg/m2
2. Cumulative anthracycline doses:

   * 125-175 mg/m2
   * 200-250 mg/m2
   * 275-325 mg/m2
   * After maximal anthracycline treatment
   * One year after completion of maximal anthracycline therapy

The blood tests being done are:

Matrix/Fibrosis pathway:Plasma levels of MMPs (all soluble MMP types) and TIMPs, (all 4 TIMPs); Inflammatory domain: cytokines (TNFα, interleukins, interferon gamma (IFNG), TGF β2, TGF βII)), Cytokine receptors (sTNF RI, sTNF RII, sSt2, sgp130, siL1- RII/sCD121b, siL-2Rα/CD25, siL-4R, siL-6R, Endoglin); Signaling pathway: growth factors (GDP-15, GCSF, VEGF, sVEGFR2 TGFβ1, IGF-1;

ELIGIBILITY:
Inclusion Criteria:

* - Age (≥9years old)
* Newly diagnosed with a malignancy that is anticipated to receive high dose anthracyclines as part of their chemotherapy (such as but not limited to solid tumors, high risk Acute Lymphocytic Leukemia, Acute myelogenous Leukemia and lymphomas)
* Parental/caregiver consent and subject assent to enrollment

Exclusion Criteria:

* - Contraindications to CMRI.*
* Patients requiring sedation for the CMRI procedure
* Pregnancy tests are done routinely prior to chemotherapy, if test is positive the patient will be excluded
* Subject is too large to be safely accommodated by MRI
* Serum creatinine higher than the guidelines for adequate renal function

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Age group is greater than or equal to 9 years of age, have a cancer diagnosis that will be treated with anthracyclines
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2013-02; Primary Completion 2016-06-24 (Actual); Study Completion 2023-06-24 (Actual)

PRIMARY OUTCOMES:
Myocardial edema | Time points will be measured over a 1 year time frame
  Myocardial edema in the acute phase measured by a composite of multiple measures that include T1 and T2 mapping, signal enhancement in T2 weighted images.
Regional wall motion abnormalities | Time points will be measured over a 1 year time frame
  Decrease in myocardial strain and strain rate compared to baseline calculations
Biomarkers of adverse cardiac remodeling | Time points will be measured over a 1 year time frame
  Elevation of serologic biomarkers CRP, Troponin, Caspases, BNP, and extracellular matrix remodeling (PCIP, CITP, PICP/CITP ratio, MMPs and MMPs/TIMP ratio

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Berthod (Ruiz), MSN, RN, CPN, CCRC, Principal Investigator — Connecticut Childrens Medical Center
Locations (1):
- Olga H Toro-Salazar, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Toro-Salazar OH, Lee JH, Zellars KN, Perreault PE, Mason KC, Wang Z, Hor KN, Gillan E, Zeiss CJ, Gatti DM, Davey BT, Kutty S, Liang BT, Spinale FG. Use of integrated imaging and serum biomarker profiles to identify subclinical dysfunction in pediatric cancer patients treated with anthracyclines. Cardiooncology. 2018;4:4. doi: 10.1186/s40959-018-0030-5. Epub 2018 May 1. PMID 29900007